CLINICAL TRIAL: NCT06132750
Title: A 5-year Natural History Study in LAMA2-related Muscular Dystrophy and SELENON-related Myopathy: the Extended LAST STRONG Study
Brief Title: A 5-year Natural History Study in LAMA2-related Muscular Dystrophy and SELENON-related Myopathy.
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84381.091.23
Record Dates: First submitted 2023-10-05; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: LAMA2-related Muscular Dystrophy; SELENON-related Myopathy
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SELENON-related myopathy or LAMA2-related muscular dystrophy: Participants diagnosed with congenital myopathy/muscular dystrophy due to mutations in the SEPN1 (SELENON) or LAMA2 gene
  Interventions: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
SELENON-related myopathy (SELENON-RM) and LAMA2-related muscular dystrophy (LAMA2-MD) are congenital neuromuscular disorders presenting with slowly, progressive axial muscle weakness, spinal rigidity, scoliosis and respiratory insufficiency. Currently, no curative treatment options exist, yet promising preclinical trials are ongoing. Clinical trials are expected to start within 5 years. Natural history data and outcome measures for measuring therapy effectiveness were lacking. Therefore, the LAST STRONG Study (a 1.5-year natural history study) started in 2020. With the extended LAST STRONG Study, we aim to further analyze and expand the 1.5-year natural history data on SELENON-RM or LAMA2-MD to provide a detailed clinical description of the Dutch and Flemish cohort. This will enable a smooth transition towards implementation into clinical care and clinical trials.

The extended LAST STRONG Study is a prospective, observational natural history study in Dutch-speaking patients of all ages diagnosed with SELENON-RM and LAMA2-MD. Patients will be invited to visit our hospital two times (3- and 5-years) after the first visit in the LAST STRONG Study. During both visits, patients will undergo a subset of tests (neurological examination, functional measurements, questionnaires, muscle ultrasound, MRI, pulmonary assessment and accelerometry). All measurements are adapted to the patient's age and functional disabilities.

DETAILED DESCRIPTION:
Rationale: A long-term prospective natural history study in an unselected group of patients including clinical and functional outcome measures is lacking in both SELENON-related myopathy (SELENON-RM) and LAMA2-related muscular dystrophy (LAMA2-MD). Due to the promising ongoing preclinical trials, there is a high need to obtain natural history data in order to reach trial readiness for both diseases. With the extended LAST STRONG study, we aim to further analyze and expand our 1.5-year natural history data on SELENON-RM and LAMA2-MD to provide a detailed clinical description of the Dutch and Flemish cohort. This will enable a smooth transition towards implementation into clinical care and clinical trials that are expected to start within 5 years.

Objective: (1) To collect 3- and 5-year natural history data in patients with SELENON-RM and LAMA2-MD. (2) Implementation of natural history data collection into clinical care and international guidelines, and reach trial readiness.

Study design: This is an observational study. A variety of tests will be performed to get a full impression of the patient's abilities and disabilities (standard medical history, neurological examination, functional measurements, questionnaires, imaging, pulmonary assessment and accelerometry). The tests that the patient undergoes depend on the age/abilities/wishes. The tests are selected based on our previously performed 1.5-year natural history study in LAMA2-MD and SELENON-RM. Each participant will perform these measurements during the two scheduled visits at 3- and 5-year after the first visit during the LAST STRONG Study.

Risk and benefit assessment: This study does not concern any product (medicinal product, food product or medical device). There is a small risk for minor injury, e.g. when a participant falls. However since the investigators use all functional tests using movements to which most participants are familiar (i.e. walking, transfers, etc.), the participant will be able to estimate his/her own risk. The investigators don't include tests in which they push participants to their physical limits. the investigators conclude that this study has a negligible risk. A benefit includes the possibility for participants to get a detailed analysis on their own health. Additionally, participants will contribute to the design of future clinical trials on possible treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to complete (part of) the measurement protocol at the Radboudumc, Nijmegen. If patients do not wish or not able to visit our neuromuscular center, they are offered to participate in our study through home visits.
* Genetic conformation of LAMA2-related muscular dystrophy or SELENON-related myopathy by two recessive (likely) pathologic mutations in the LAMA2 or SELENON gene.
* Typical clinical and histological characteristics combined with genetic confirmation in a first degree relative.
* Dutch speaking

Exclusion Criteria:

* Insufficient understanding of the Dutch language

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SELENON-RM patients (prevalence: 0.5 in 1.000.000) and LAMA2-RM patients (prevalence: 4 in 500.000) are rare and no Dutch registry exists. Therefore, the investigators can only estimate the number of patients in the Netherlands and Belgium. All patients with SELENON-RM and LAMA2-MD mutations will be identified through contact with genetic diagnostic services, rehabilitation centers, and muscle disease experts in The Netherlands and Dutch-speaking Belgium.
  In the LAST STRONG Study, 27 LAMA2-MD patients (21±13 years) and 11 SELENON-RM (20±13 years) patients were included. Based on this high participation rate and the minimal loss from follow-up, we expect between 35 to 40 patients to participate in the extended LAST STRONG Study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of Motor Function Measure (MFM)-32 (older than 7 years) of MFM-20 (2 to 7 years old) | Change from baseline to 3 years and 5 years
  Global motor functioning. The items of the MFM are classified in 3 domains: D1: standing and transfers, D2: Axial and proximal motor function, D3: Distal motor function. Higher scored indicate a better outcome. The range of the total score is 0-96. The main point of interest includes the change of MFM score over a period of 5 years.

SECONDARY OUTCOMES:
Change of physical activity in daily life assessed by an accelerometer (GENEActiv original devices) for 7 days | Change from baseline to 3 years and 5 years
  Physical activity in daily life will be assessed by wearing an accelerometer (GENEActiv original devices) for 7 days.
Change of activity limitations assessed using ACTIVLIM (6 years and older) | Change from baseline at 3 years and 5 years
  ACTIVLIM assesses the ability to perform 22 activities of daily life on a 3-point scale from impossible to easy.
Change of bone density assessed using DEXA-scan (2 years and older) | Change from baseline at 3 years and 5 years
  The bone density of the spine and hip will be measured by a DEXA scan.
Change of The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) score (children under the age of 2 years) | Change from baseline at 3 years and 5 years
  CHOP INTEND assesses motor skills of children below 2 years of age.
Change of fatigue (pediatric 2-17 years old) assessed by PedsQL Multidimensional Fatigue Scale (MFS) | Change from baseline at 3 years and 5 years
  PedsQL MFS assesses subjective fatigue in three domains.
Change of functional ability in daily life assessed by Egen klassification scale version 2 (EK2) (16 years and older) | Change from baseline at 3 years and 5 years
  The EK2 is a questionnaire that was designed to measure functional ability of activities in daily living in non-ambulant Duchenne muscular dystrophy patients. This questionnaire is only available in English. Therefore, only participants of 16 years and older who have a sufficient understanding of the English language will be asked to complete this questionnaire.
Change of Functional Ambulation Category (FAC) (5 years and older) | Change from baseline at 3 years and 5 years
  The FAC assesses functional ambulation in participants.
Change of Graded and Timed function tests | Change from baseline at 3 years and 5 years
  The time (in sec) it takes to complete functions of the lower extremity will be assessed with the 30 seconds sit to stand test, the time it takes to climb 4 stairs, the time it takes to descend 4 stairs and the time it takes to rise from the floor.
Change of Hammersmith Infant Neurological Examination (HINE) (under the age of 2 years) | Change from baseline at 3 years and 5 years
  HINE is designed to be a simple and scorable method for evaluating infants from 2 months to 2 years of age. It includes three sections that assess different aspects of neurologic function, including neurological examination, developmental milestones and behavioral assessment.
Change of Impact on Participation and Autonomy (IPA) (18 years and older) | Change from baseline at 3 years and 5 years
  Questionnaire about participation and autonomy in daily life.
Change of maximal voluntary isometric contraction (5 years and older) | Change from baseline at 3 years and 5 years
  Maximal voluntary isometric contraction will be measured by hand-held dynamometry.
Change of location, level and characteristics of pain assessed by McGill pain questionnaire (12 years and older) | Change from baseline at 3 years and 5 years
  Questionnaire in which the location, level and characteristics of pain are assessed.
Change of muscle atrophy (cm) assessed by muscle ultrasound | Change from baseline at 3 years and 5 years
  Muscle atrophy of the leg, arm and abdominal muscles will be assessed by muscle ultrasound.
Change of muscle fattening (echo-intensity) assessed by muscle ultrasound | Change from baseline at 3 years and 5 years
  Muscle fattening of the leg, arm and abdominal muscles will be assessed by muscle ultrasound.
Change of muscle fattening by quantitative lower extremity muscle MRI (10 years and older) | Change from baseline at 3 years and 5 years
  A lower extremity MRI will be performed in participants who are able to lie supine and still for 20 minutes and who are not dependent on respiratory equipment. Muscle fattening will be assessed by Regions of interest (ROIs) and modified Mercuri score.
Change of muscle atrophy by quantitative lower extremity muscle MRI (10 years and older) | Change from baseline at 3 years and 5 years
  A lower extremity MRI will be performed in participants who are able to lie supine and still for 20 minutes and who are not dependent on respiratory equipment. Muscle atrophy will be assessed by muscle volume score.
Change of muscle power assessed by muscle power measurements (Medical Research Council (MRC) scale) (2 years and older) | Change from baseline at 3 years and 5 years
  Muscle power of individual muscle groups can be assessed by muscle power measurements and graded in correspondence with the MRC scale.
Pulmonary function (5 years and older) - change of forced vital capacity (percentage predicted) | Change from baseline at 3 years and 5 years
  Obtained with handheld spirometry in sit and supine.
Pulmonary function (5 years and older) - change of forced expiratory volume in the first second (liter) (percentage predicted) | Change from baseline at 3 years and 5 years
  Obtained with handheld spirometry in sit and supine
Pulmonary function (5 years and older) - change of peak expiratory flow (liter per second) | Change from baseline at 3 years and 5 years
  Obtained with handheld spirometry in sit and supine
Pulmonary function (5 years and older) - change of vital capacity (percentage predicted) | Change from baseline at 3 years and 5 years
  Obtained with handheld spirometry in sit and supine
Pulmonary function (5 years and older) - change of peak cough flow (liter per second) | Change from baseline at 3 years and 5 years
  Obtained with handheld spirometry in sit and supine
Pulmonary function (5 years and older) - change of maximal expiratory pressure (cmH2O) | Change from baseline at 3 years and 5 years
  Obtained with handheld device
Pulmonary function (5 years and older) - change of maximal inspiratory pressure (cmH2O) | Change from baseline at 3 years and 5 years
  Obtained with handheld device
Pulmonary function (5 years and older) - change of sniff nasal inspiratory pressure (cmH2O) | Change from baseline at 3 years and 5 years
  Obtained with handheld device
Change of Quality of life (adult) assessed by SF36/RAND36 | Change from baseline at 3 years and 5 years
  The Quality of Life is measured by the SF36/RAND36 questionnaire. This questionnaire addresses eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a singe item that provides an indication of perceived change in health.
Change of Quality of Life (adult) assessed by Individualized Neuromuscular Quality of Life (INQoL) | Change from baseline at 3 years and 5 years
  The INQoL is a validated muscle disease specific measure of quality of life, which can be used for individuals or large samples.
Change of Quality of Life (pediatric; 2-17 years old) assessed by PedsQL neuromuscular module (NMM) | Change from baseline at 3 years and 5 years
  The PedsQL NMM questionnaire consists of 25 questions in three domains: Neuromuscular disease, communication and family resources.
Change of range of motion of elbows, wrist, hips, knee and ankle | Change from baseline at 3 years and 5 years
  The range of motion of elbows, wrist, hips, knee and ankle is noted bilaterally by goniometry.
Change of Brooke and Vignos scale (2 years and older) | Change from baseline at 3 years and 5 years
  The Brooke and Vignos scale provide ordinal data to assess the upper and lower extremity functions.
Change of Wong-Baker Faces Pain Scale (2 years and older) | Change from baseline at 3 years and 5 years
  The Wong-Baker Faces Pain Scale was originally created for children to help them communicate about their pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Research data is open access shared upon publication, provided that this complies with privacy regulations. The Donders Repository is the default repository for sharing the investigators' data.

REFERENCES:
- [Derived] de Laat ECM, Houwen-van Opstal SLS, Bouman K, van Doorn JLM, Cameron D, van Alfen N, Dittrich ATM, Kamsteeg EJ, Smeets HJM, Groothuis JT, Erasmus CE, Voermans NC. A 5-year natural history study in LAMA2-related muscular dystrophy and SELENON-related myopathy: the Extended LAST STRONG study. BMC Neurol. 2024 Oct 23;24(1):409. doi: 10.1186/s12883-024-03852-4. PMID 39443859